CLINICAL TRIAL: NCT04280003
Title: Allogeneic Adipose Tissue-derived Mesenchymal Stem Cells in Ischemic Stroke. A Phase IIB Multicenter Double Blind Placebo Controlled Clinical Trial
Brief Title: Allogeneic Adipose Tissue-derived Mesenchymal Stem Cells in Ischemic Stroke
Acronym: AMASCIS-02
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMASCIS - 02
Record Dates: First submitted 2019-08-06; First posted 2020-02-21 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2022-05

CONDITIONS: Ischemic Stroke; Adipose Tissue-derived Stem Cell; Functional Status
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Two different treatment grupos; intravenous alogenic adipose tissue-derived mesenchymal stem cells or intravenous placebo solution
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment and placebo solutions have identical appearance. Protocols will be designed to ensure that the physician evaluating patient safety and efficacy outcome as well as laboratory analysis, will not have access to the randomisation codes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): 15 patients will receive intravenous alogenic adipose tissue-derived stem cells in a single dose of one million cells per kg.
  Interventions: Other: Alogenic adipose tissue-derived stem cells
- Placebo group (Placebo Comparator): 15 patients will receive a single intravenous placebo solution with the same appearance as the treatment group.
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Other: Alogenic adipose tissue-derived stem cells — Concentration of the cells: 10 million cells / ml
  Arms: Treatment group
Drug: Placebo solution — Placebo intravenous solution, same appearance stem cells solution
  Arms: Placebo group

SUMMARY:
This is a multicenter, doble blind, placebo controlled clinical trial to asses de safety and efficacy of intravenous administration of alogenic adipose tissue-derived mesenchymal stem cells in the first four days from acute ischemic stroke.

DETAILED DESCRIPTION:
Two spanish hospitals with teams experienced in stroke management will participate in this study, recruiting a total of 30 patients between them both. After confirming that patients fulfill the inclusion criteria and none of the exclusion criteria, informed consent will be signed and randomization will take place (1:1). There are two different groups of treatment; the first group will be treated with intravenous alogenic adipose tissue-derived stem cells (at a concentration of one million cells per kg) within the first four days from stroke onset, the second group will be treated will an intravenous placebo solution. Follow-up will last for 24 months during which safety issues such as adverse events and neurological and systemic complications will be assessed at 24 hours, 7 days and 3, 6, 12,18 and 24 months after treatment. Neurological disability using the modified Rankin Scale and National Institute of Health Stroke Scale will also be registered in every scheduled visit. Biochemical markers of tissue repair (GM-CSF, BDNF, VEGF, TGF-1, GFAP, MBP, MMP-3) as well as extracellular vesicles will be extracted on baseline visit as well as 7 days and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke patients > 18 years old
* Patients must be able to be treated within the first 4 days (+/- 1) from acute stroke symptoms onset. If the time of symptom onset is unknown, this shall refer to the last time the patient was observed as asymptomatic.
* A computed tomography (CT) or magnetic resonance imaging (MRI) scan compatible with the clinical diagnosis of acute non-lacunar IS in the region of the middle cerebral artery (with cortical or subcortical involvement).
* A score on the National Institute of Health Stroke Scale (NIHSS) of 8-20, with at least two of these points in sections 5 and 6 (motor deficit) at the time of inclusion. NIHSS evaluation for screening of these patients will take place after finalization of reperfusion therapies (if they have been performed) providing that the clinical condition of the patient is stable with no prevision of immediate recovery. A measurable focal neurologic disabilty must persist to the time of treatment.
* A prestroke score on the Modified Rankin Scale (mRS) ≤1 (no significant disability).
* Female subjects non-child bearing potential. Female subjects who are of non-childbearing potential are defined as meeting at least 1 of the following criteria:

Have undergone a documented hysterectomy and/or bilateral oophorectomy; Have medically confirmed ovarian failure; or Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause.

* Female subjects of child-bearing potential need a negative pregnancy test and must agree to use adequate contraception for the duration of the study (from screening through the final of the study). The following types of contraception are considered adequate provided they are locally authorized for use: oral, transdermal, or injectable (depot) estrogen and/or progestogen, selective estrogen receptor modulator therapy, intrauterine contraceptive device, double barrier method (e.g., condom and diaphragm or spermicidal gel) or vasectomy.
* Signed informed consent

Exclusion Criteria:

* Comatose patients; patients with a score of 2 or more on item 1a of the NIHSS related to the degree of awareness.
* Evidence on neuroimaging of brain tumour, cerebral oedema with midline shift and a clinically significant compression of ventricles, cerebellar or brainstem infarction and intraventricular, intracerebral or subarachnoid haemorrhage. Small petechial haemorrhages are not exclusion criteria.
* Current drug or alcohol use or dependence
* Active infectious disease, including human immunodeficiency virus, hepatitis B, and hepatitis C. A controlled infection is not an exclusion criterion.
* Pre-existing dementia.
* A health status, any clinical condition (eg, short life expectancy, and coexisting disease or a surgical or endovascular planned procedure) or other characteristic that precludes appropriate diagnosis, treatment, or follow-up in the trial.
* Patients who are participating in another clinical trial.
* Inability or unwillingness of the individual or their legal guardian/representative to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Safety of administration of adipose tissue-derived mesenchymal stem cells measured as reported adverse events | Up to 24 months after treatment or placebo administration
  Adverse events reported spontaneously or in response to questions not addressed.
Safety of administration of adipose tissue-derived mesenchymal stem cells measured as neurological o systemic complications | Up to 24 months after treatment or placebo administration
  Neurological or systemic complications

SECONDARY OUTCOMES:
Efficacy of administration of adipose tissue-derived mesenchymal stem cells measured by the Modified Rankin Scale | Up to 24 months after treatment or placebo administration
  Modified Rankin Scale (mRS): success is considered when the patient obtains a score of 0-3, and failure include scores of 4 to 6 at months 3,6,12 and 24. An additional exploratorry efficacy analysis of mRS shift at months 3,6,12 and 24 will also be made.
Efficacy of administration of adipose tissue-derived mesenchymal stem cells measured by the NIHSS | Up to 24 months after treatment or placebo administration
  National Institute of Health Stroke Scale. It will be measured at all scheluded visits. Success is defined as an improvement of 75% or more from baseline. An additional exploratory analysis will look for differences in the distribution of median (IQR) and in the frequency of NIHSS ≤ 1between groups.
Efficacy of administration of adipose tissue-derived mesenchymal stem cells measuring blood brain repair biomarkers | Up to 3 months after treatment or placebo administration
  Brain repair biomarkers in blood samples (GM-CSF, PDGF-BB, BDNF, VEGF, TGF-1, GFAP, MBP, MMP-3 and extracelular vesicles) measured at baseline, day 7 and mnth 3 after treatment or placebo administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be available from the corresponding author on reasonable request, considered compliant General Data Protection Regulation and the data-sharing agreement is approved by the relevant Spanish authorities. Upon study finalization, anonymized individual patient data will be available on a public repertoire of the Community of Madrid.

REFERENCES:
- [Background] de Celis-Ruiz E, Fuentes B, Moniche F, Montaner J, Borobia AM, Gutierrez-Fernandez M, Diez-Tejedor E. Allogeneic adipose tissue-derived mesenchymal stem cells in ischaemic stroke (AMASCIS-02): a phase IIb, multicentre, double-blind, placebo-controlled clinical trial protocol. BMJ Open. 2021 Aug 9;11(8):e051790. doi: 10.1136/bmjopen-2021-051790. PMID 34373315